CLINICAL TRIAL: NCT05946382
Title: A Comparison of Two Ultra-brief Interventions in Primary Care for Patients With Anxiety, Depression, and Stress: a Randomized Controlled Trial.
Brief Title: A Comparison of Two Ultra-brief Interventions in Primary Care for Patients With Anxiety, Depression, and Stress.
Acronym: RNTACTSweden
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-06465-01
Record Dates: First submitted 2023-06-22; First posted 2023-07-14 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Mental Disorder; Mental Health Issue; Mental Depression; Anxiety; Mental Stress; Rumination - Thoughts
MeSH Terms: conditions — Mental Disorders; Depression; Anxiety Disorders; Stress, Psychological | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: After assessment the participant receives either the RNT-ACT arm or the iCBT arm.
  When the treatment is finished, the patient is called to an evaluation visit. If the person still needs care, we are faced with two choices. Either the patient is offered usual care and is thus removed from the three-month follow-up.Or it will wait for three-month follow up.
Masking Description: Patients are made aware of the study through information material at the primary care unit in the waiting room and on the therapists door. There they can notify the contact person about their interest. Letter with information about the study will be sent out to the interested patient. If the patient chooses to participate by answering positively on the information letter, they will be contacted by telephone by a psychologist at the respective primary care unit for the opportunity to ask questions and to book an appointment for a baseline measurement at the unit. After the baseline measurement the patient is randomly assigned to one of the treatment arms. Measurements with all self-assessment scales are carried out at week 0, at the end of treatment and 3 months after the end of treatment. The participants are then offered the opportunity for a follow-up 12 months after completion of treatment using the same scales as the 3-month follow-up.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RNT-ACT protocol (Experimental): Participants randomized to RNT-ACT will receive a total of 2 sessions of 60 minutes each as well as audio files to listen to between the occasions administered via internet. Previous studies have indicated that it doesn't make much of a difference whether the temporal distance between session 1 and session 2 is between 1 week and up to 3 months. At occasion 1, the time for occasion 2 is set. The temporal distance in days will noted for each patient. The treatment is inserted into the therapist's regular diary with 60 minutes session time and appropriate break before and after the treatment (e.g. at least 5-10 minutes) for preparation and post-administration where journal writing is included.
  Interventions: Behavioral: RNT-ACT Protocol
- iCBT treatment (Active Comparator): The people randomized to Internet treatment will be offered based on M.I.N.I 7.0 a suitable iCBT program in the Stöd och Behandling (SoB) platform. The patients follow a structured self-help material which can be seen as a standard treatment option in Region Skåne, "treatment as usual". The therapist has access to the material and the patient and the therapist can communicate via a chat function. The patients are matched to iCBT programs based on whether they are most likely to show symptoms of depression or anxiety. The main component of Internet processing consists of a structured self-help program in approximately eight modules, somewhat varying depending on which program in use. The program is based on proven CBT interventions for each problem area with a strong emphasis on psychoeducation but where different intervention elements is included.
  Interventions: Behavioral: iCBT Treatment

INTERVENTIONS:
Behavioral: RNT-ACT Protocol — Swedish Translation of the 2*60 minute Acceptance and Commitment Protocol for Repetitive Negative Thinking.
  Other Names: Acceptance and Commitment Therapy (ACT)
  Arms: RNT-ACT protocol
Behavioral: iCBT Treatment — Internet-based Cognitive Behavioral Therapy as mandatory routine care in Swedish Primary care and therefore considered Treatment as usual.
  Arms: iCBT treatment

SUMMARY:
The goal of this clinical trial is to compare the effect and time consumption of the Swedish translation of the protocol for RNT-ACT with the internet administrated self-help treatment with therapist support (iCBT) for patients seeking medical care for depression, anxiety or stress at their primary care unit. The trial consists of a feasibility study and a randomized controlled trial with 3- and 12-month follow ups.

DETAILED DESCRIPTION:
The main question it aims to answer are: Is the Swedish translation of a psychological treatment protocol targeting Repetitive Negative Thinking (RNT) based on Acceptance and Commitment therapy (ACT), RNT-ACT, an effective treatment in Swedish primary care for the treatment of people with a high proportion of negative repetitive thoughts, who meet diagnostic criteria for depression and/or anxiety? The question is planned to be elaborated into the following parts:

A feasibility study in which the material and the system are tested at a single care center.

A randomized controlled trial conducted at several health centers where the comparison group is patients who are actualized for traditional psychological treatment in the form of iCBT for either anxiety or depression programs and where they are offered the second treatment arm after 3- and 12-month follow-ups.

A follow-up study where time consumption and patient satisfaction are evaluated in both branches.

Participants will be given either RNT-ACT or iCBT as treatment. The group who are given RNT-ACT will receive 2*60 minutes of therapy along with mindfulness files to listen to daily between sessions. The group who are given iCBT will receive internet-based Cognitive Behavioral Therapy, one of the forms of delivering Cognitive behavioral therapy that is implemented in Region Skåne and can thus be seen as treatment as usual. Patients will access the treatment through a secure website and communicate with their therapist by text when needed. Researchers will compare the RNT-ACT and iCBT groups to see if there are differences in depressive, anxiety- and stress- related symptoms, rumination, psychological flexibility, client satisfaction and therapist-rated time consumption. In the feasibility study researchers will also evaluate drop-out and recruitment rate.

ELIGIBILITY:
Inclusion Criteria:

* DASS-21 >25
* Ability to communicate in Swedish orally and in writing

Exclusion Criteria:

* Routine blood tests are carried out including blood count, thyroid hormone, liver status and fluid balance in order to be able to differentially diagnose any physical illness.

In addition to physical illness are exclusion criteria

* Other psychological or psychiatric treatment,
* Suicidality, substance abuse, Anorexia Nervosa, psychosis, bipolar disorder, attention deficit hyperactivity disorder (ADHD) and antisocial personality disorder (as verified based on M.I.N.I 7.0).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
DASS-21 | From assessment to 3 month follow up.
  Depression, Anxiety and Stress Scale-21 (DASS-21); Min 0, Max 63 with high values associated with more Depression/Anxiety/Stress.

SECONDARY OUTCOMES:
Drop Out rate | Up to three months.
  Percentage of patients who for any reason fails to continue in the trial until the end of intervention.
Recruitment rate | one month.
  How many patients were recruited on average for one month in the primary care unit responsible for the feasibility study.
CSQ-8 | From assessment to 3 month follow up.
  Client Satisfaction Questionnaire (CSQ-8). Min 8, Max 32 with higher values indicating higher satisfaction.
Self registered time consumption | Up to three months.
  Self-registered time consumption for therapists.
WAI | From assessment to 3 month follow up.
  Working Alliance Inventory (WAI). Min 7, Max 84 with higher values indicating better working alliance.
RRS-BR | From assessment to 3 month follow up.
  Ruminative Responses Scale - Brooding and Reflection (RRS-BR). Min 5, Max 20. A higher value indicates a higher extent of ruminative response style and self-reflection.
BSRI | From assessment to 3 month follow up.
  Brief State Rumination Inventory (BSRI). Min 0, Max 80. A higher value indicates higher degree of ongoing ruminative cognitive responses.
SAAQ | From assessment to 3 month follow up.
  Swedish Acceptance and Action Questionnaire (SAAQ). Min 6, Max 42. A higher value indicates lower psychological flexibility which indicates a worse value.
AFQ-Y8 | From assessment to 3 month follow up.
  Avoidance and Fusion Questionnaire for Youth (AFQ-Y8). Min 0, Max 32. A higher value indicates lower psychological flexibility which indicates a worse value.
CFQ-7 | From assessment to 3 month follow up.
  Cognitive Fusion Questionnaire - 7 items (CFQ-7). Min 1, Max 49. A higher value indicates higher cognitive fusion which indicates a worse value.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Milos Nymberg, PhD, Principal Investigator — Lund University/Region Skåne
Locations (1):
- Vårdcentralen Laröd, Helsingborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alfonsson S, Wallin E, Maathz P. Factor structure and validity of the Depression, Anxiety and Stress Scale-21 in Swedish translation. J Psychiatr Ment Health Nurs. 2017 Mar;24(2-3):154-162. doi: 10.1111/jpm.12363. Epub 2017 Jan 25. PMID 28124410
- [Background] Amorim P, Lecrubier Y, Weiller E, Hergueta T, Sheehan D. DSM-IH-R Psychotic Disorders: procedural validity of the Mini International Neuropsychiatric Interview (MINI). Concordance and causes for discordance with the CIDI. Eur Psychiatry. 1998;13(1):26-34. doi: 10.1016/S0924-9338(97)86748-X. PMID 19698595
- [Background] Andersson G, Titov N, Dear BF, Rozental A, Carlbring P. Internet-delivered psychological treatments: from innovation to implementation. World Psychiatry. 2019 Feb;18(1):20-28. doi: 10.1002/wps.20610. PMID 30600624
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Berger T, Urech A, Krieger T, Stolz T, Schulz A, Vincent A, Moser CT, Moritz S, Meyer B. Effects of a transdiagnostic unguided Internet intervention ('velibra') for anxiety disorders in primary care: results of a randomized controlled trial. Psychol Med. 2017 Jan;47(1):67-80. doi: 10.1017/S0033291716002270. Epub 2016 Sep 22. PMID 27655039
- [Background] Donati MA, Berrocal C, Bernini O, Gori C, Primi C. Measuring cognitive fusion through the Cognitive Fusion Questionnaire-7: Measurement invariance across non-clinical and clinical psychological samples. PLoS One. 2021 Feb 3;16(2):e0246434. doi: 10.1371/journal.pone.0246434. eCollection 2021. PMID 33534868
- [Background] Gillanders DT, Bolderston H, Bond FW, Dempster M, Flaxman PE, Campbell L, Kerr S, Tansey L, Noel P, Ferenbach C, Masley S, Roach L, Lloyd J, May L, Clarke S, Remington B. The development and initial validation of the cognitive fusion questionnaire. Behav Ther. 2014 Jan;45(1):83-101. doi: 10.1016/j.beth.2013.09.001. Epub 2013 Sep 18. PMID 24411117
- [Background] Glasgow RE, Fisher L, Strycker LA, Hessler D, Toobert DJ, King DK, Jacobs T. Minimal intervention needed for change: definition, use, and value for improving health and health research. Transl Behav Med. 2014 Mar;4(1):26-33. doi: 10.1007/s13142-013-0232-1. PMID 24653774
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Lundgren T, Parling T. Swedish Acceptance and Action Questionnaire (SAAQ): a psychometric evaluation. Cogn Behav Ther. 2017 Jun;46(4):315-326. doi: 10.1080/16506073.2016.1250228. Epub 2016 Dec 9. PMID 27931161
- [Background] Ruiz FJ, Pena-Vargas A, Ramirez ES, Suarez-Falcon JC, Garcia-Martin MB, Garcia-Beltran DM, Henao AM, Monroy-Cifuentes A, Sanchez PD. Efficacy of a two-session repetitive negative thinking-focused acceptance and commitment therapy (ACT) protocol for depression and generalized anxiety disorder: A randomized waitlist control trial. Psychotherapy (Chic). 2020 Sep;57(3):444-456. doi: 10.1037/pst0000273. Epub 2020 Jan 16. PMID 31944806
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Ehring, T., & Watkins, E. R. (2008). Repetitive negative thinking as a transdiagnostic process. International Journal of Cognitive Therapy, 1(3), 192-205. https://doi.org/10.1521/ijct.2008.1.3.192
- [Background] Horvath, A. O., & Greenberg, L. S. (1989). Development and validation of the Working Alliance Inventory. Journal of Counseling Psychology, 36(2), 223-233. https://doi.org/10.1037/0022-0167.36.2.223
- [Background] Livheim, F., Tengström, A., Bond, F. W., Andersson, G., Dahl, J., & Rosendahl, I. (2016). Psychometric properties of the Avoidance and Fusion Questionnaire for Youth: A psychological measure of psychological inflexibility in youth. Journal of Contextual Behavioral Science, 5(2), 103-110. https://doi.org/10.1016/j.jcbs.2016.04.001
- [Background] Lecrubier, Y., Sheehan, D., Weiller, E., Amorim, P., Bonora, I., Sheehan, K., . . . Dunbar, G. (1997). The Mini International Neuropsychiatric Interview (MINI). A short diagnostic structured interview: Reliability and validity according to the CIDI. European Psychiatry, 12(5), 224-231. doi:10.1016/S0924-9338(97)83296-8
- [Background] Marchetti, I., Mor, N., Chiorri, C. et al. The Brief State Rumination Inventory (BSRI): Validation and Psychometric Evaluation. Cogn Ther Res 42, 447-460 (2018). https://doi.org/10.1007/s10608-018-9901-1
- [Background] O'Neill, L., Latchford, G., McCracken, L. M., & Graham, C. D. (2019). The development of the acceptance and commitment therapy fidelity measure (ACT-FM): A Delphi Study and field test. Journal of Contextual Behavioral Science, 14, 111-118. https://doi.org/10.1016/j.jcbs.2019.08.008
- [Background] Schermuly-Haupt, ML., Linden, M. & Rush, A.J. Unwanted Events and Side Effects in Cognitive Behavior Therapy. Cogn Ther Res 42, 219-229 (2018). https://doi.org/10.1007/s10608-018-9904-y
- [Background] Treynor, W., Gonzalez, R. & Nolen-Hoeksema, S. Rumination Reconsidered: A Psychometric Analysis. Cognitive Therapy and Research 27, 247-259 (2003). https://doi.org/10.1023/A:1023910315561
- [Background] Silberleitner, N., Cederwald, A. von, & Robinson, P. (2021). Integrerad primärvård: Principer, färdigheter och rutiner för hela vårdcentralens arbete med Beteenderelaterad Ohälsa. Natur & Kultur.
- See also: Client Satisfaction Questionnaire scales — https://csqscales.com/
- See also: Swedish platform for use of internet service in health care — https://www.inera.se/tjanster/alla-tjanster-a-o/stod-och-behandling/
- See also: Social Psychology Network. Research randomizer. — https://www.randomizer.org/
- See also: Swedish authority (Socialstyrelsen). April 2021. National guidelines for care in depression and anxiety disorders. Support for governance and management. — https://www.socialstyrelsen.se/globalassets/sharepoint-dokument/artikelkatalog/nationella-riktlinjer/2021-4-7339.pdf
- See also: Swedish authority (Socialstyrelsen) February 2018. Accessibility in health and healthcare — https://www.socialstyrelsen.se/globalassets/sharepoint-dokument/artikelkatalog/ovrigt/2018-2-16.pdf
- See also: Working Alliance Inventory. — https://wai.profhorvath.com/downloads
- See also: The Swedish governments official investigations. Statens Offentliga Utredningar (SOU) 2021:6 Good and close care - The right support for mental health — https://www.regeringen.se/rattsliga-dokument/statens-offentliga-utredningar/2021/01/sou-20216/
- See also: State of the act evidence | association for contextual behavioral science. — https://contextualscience.org/state_of_the_act_evidence